CLINICAL TRIAL: NCT05708976
Title: HypErthermia as an Additional Treatment for the Biology and Experience of Depression: Study 2
Acronym: HEATBED2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-34246; R34AT011221 (NIH)
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Depression
Keywords: hyperthermia; heat therapy; passive heating
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Hyperthermia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two study arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Study clinicians, who perform clinical interviews and provide cognitive behavioral therapy (CBT) treatments, will be masked to participant condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Whole-body Hyperthermia (Active Treatment) (Experimental): Participants receive 8 cognitive behavioral therapy (CBT) sessions and 4 bi-weekly whole-body hyperthermia (WBH) sessions that raise core body temperature to 38.5 C. Each active WBH session (including preparation and post-session activities) is up to approximately 3.5 hours, and each CBT session is approximately 50 minutes.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Device: Active Whole-Body Hyperthermia (Active WBH)
- Sham Whole-body Hyperthermia (Sham Treatment) (Placebo Comparator): Participants receive 8 cognitive behavioral therapy (CBT) sessions and 4 bi-weekly sham whole-body hyperthermia (WBH) sessions, which minimally raise body temperature. Each sham WBH session (including preparation and post-session activities) is up to approximately 3.5 hours, and each CBT session is approximately 50 minutes.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Device: Sham Whole-Body Hyperthermia (Sham WBH)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy (CBT) is a behavioral (psychotherapeutic) intervention for major depressive disorder (MDD). A highly trained masters' or PhD-level clinician will administer 8 weekly CBT sessions (~50 minutes each), following the standard cognitive behavioral therapy for depression protocol.
Device: Active Whole-Body Hyperthermia (Active WBH) — Active whole-body hyperthermia (active WBH) will be administered by trained research assistants. Preparation for the active WBH session, the active WBH session, and cool down will last 3.5 hours, with heating lasting approximately 90-100 minutes (and no longer than 140 minutes). The treatment will take place in an infrared sauna dome, and the active heating phase will last until the participants has achieved a core (rectal) temperature of 38.5 C.
  Other Names: Active Sauna Sessions
  Arms: Active Whole-body Hyperthermia (Active Treatment)
Device: Sham Whole-Body Hyperthermia (Sham WBH) — Sham whole-body hyperthermia (sham WBH) will be administered by trained research assistants. Preparation for the sham WBH session, the sham WBH session, and cool down will last 3.5 hours, with heating lasting approximately 90-100 minutes (and no longer than 140 minutes). The treatment will take place in an infrared sauna dome, and the sham WBH session will minimally impact core body temperature.
  Other Names: Sham Sauna Sessions
  Arms: Sham Whole-body Hyperthermia (Sham Treatment)

SUMMARY:
This randomized two-arm intervention trial administers 8 weekly cognitive behavioral therapy (CBT) sessions and 4 bi-weekly active whole-body hyperthermia (active WBH) sessions or 4 bi-weekly sham WBH sessions to adults aged 18 years or older with major depressive disorder (MDD).

DETAILED DESCRIPTION:
Major Depressive Disorder afflicts more than 300 million people worldwide and is the leading cause of life years lost to disability. Current treatments have important limitations in efficacy and, in the case of medication, substantial side-effects. There is thus a compelling need for additional effective, well-tolerated treatments. One such potential treatment is whole-body hyperthermia (WBH). The investigators hypothesize that active WBH may be particularly effective in combination with cognitive behavioral therapy (CBT), an established treatment for depression. This randomized two-arm trial will pilot and optimize procedures for randomizing participants to receive CBT (8 weekly sessions) and 4 bi-weekly whole-body hyperthermia (active WBH) or 4 bi-weekly sham WBH sessions. This work holds important promise to improve treatment of depression and advance understanding of the role of integrated mind-body therapies for mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years old
* Current major depressive episode of at least 2 weeks duration as assessed by the Structured Clinical Interview for DSM-5 (SCID) and a Beck Depression Inventory-II (BDIII) score > 21 at screening
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures
* Must have smartphone onto which the participant can download an app from Apple App or Google Play stores
* Ability to lie supine (on back) for 2 hours (required for sauna sessions)

Exclusion Criteria:

* >30% reduction in BDI-II score between Screen #1 and Screen #2 (conducted ~1 week after Screen #1)
* Suicide attempt in the past 12 months defined using the SAMHSA suicidality question during the clinician-administered interview or active suicidal ideation as indexed by a score of 3 on the BDI-II suicidality item during the clinician-administered interview
* Any of the following medical conditions: cardiovascular disease (other than controlled hypertension), seizure disorder, history of cerebrovascular accident (CVA) or other serious neurological condition (e.g. Parkinson's disease, multiple sclerosis, or dementia), current neoplasia, any active enclosed infection (e.g. dental abscess, joint infection), hemophilia or other cause for excessive bleeding (e.g. platelet disorder), or other medical condition that in the opinion of investigators may increase the risk of WBH
* Comorbid psychiatric conditions or history of comorbid psychiatric conditions that might better explain depressive symptoms, including schizophrenia, schizoaffective disorder, Bipolar Disorder I, Obsessive Compulsive Disorder, Anorexia Nervosa, Bulimia Nervosa, Alcohol Dependence, or Drug Dependence
* Known hypersensitivity to hyperthermia and/or infrared exposure
* Inability to fit into the sauna device
* Breast implants
* Pregnancy, active lactation or intention to become pregnant during the study period
* Use of any medication that might impact thermoregulatory capacity, including: Diuretics, barbiturates, beta-blockers, antipsychotic agents, anti-cholinergic agents or chronic use of antihistamines, aspirin (other than low-dose ASA for prophylactic purposes), medication prescribed for the treatment of depression (antidepressant medication [ADM]) including but not limited to: selective serotonin reuptake inhibitors [SSRIs], Serotonin and norepinephrine reuptake inhibitors [SNRIs], Monoamine oxidase inhibitors [MAOIs], Tricyclics [TCAs], and atypical antipsychotic and antidepressant medications (participants must have been free of these medications for at least 4 weeks), antibiotics (past 14 days), pain medication (opioids) due to procedure, e.g., dental procedure (past 14 days), Emergency contraception pill (past 14 days) any other medication that in the judgment of the PI would increase risk of study participation or introduce excessive variance into physiological or behavioral responses to WBH recent use (multiple consecutive doses) of: non-steroidal anti-inflammatory drugs (NSAIDs), systemic corticosteroids, cytokine antagonists
* Regular use of any nicotine products, including cigarettes, vapes, chewing tobacco, or other forms of nicotine (if use is not regular, must be willing to refrain for 24 hours before and 24 hours after WBH session)
* Unwilling to refrain from using marijuana products and alcohol for the 24 hours before and 24 hours after WBH session
* Unwilling to refrain from heavy exercise on the day of WBH sessions
* Unwilling to refrain from engaging with sauna, hot yoga, cold plunges, cryotherapy, and hot tub/jacuzzi outside of study (prospective participant must not have engaged with any of these activities for 30 days prior to their baseline study visit).
* Has begun new psychotherapy treatment in the prior 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Mason, PhD, Principal Investigator — University of California, San Francisco; Frederick M Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mason AE, Fisher SM, Chowdhary A, Guvva E, Veasna D, Floyd E, Fender SB, Raison C. Feasibility and acceptability of a Whole-Body hyperthermia (WBH) protocol. Int J Hyperthermia. 2021;38(1):1529-1535. doi: 10.1080/02656736.2021.1991010. PMID 34674592
- [Background] Janssen CW, Lowry CA, Mehl MR, Allen JJ, Kelly KL, Gartner DE, Medrano A, Begay TK, Rentscher K, White JJ, Fridman A, Roberts LJ, Robbins ML, Hanusch KU, Cole SP, Raison CL. Whole-Body Hyperthermia for the Treatment of Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):789-95. doi: 10.1001/jamapsychiatry.2016.1031. PMID 27172277
- [Background] Hanusch KU, Janssen CH, Billheimer D, Jenkins I, Spurgeon E, Lowry CA, Raison CL. Whole-body hyperthermia for the treatment of major depression: associations with thermoregulatory cooling. Am J Psychiatry. 2013 Jul;170(7):802-4. doi: 10.1176/appi.ajp.2013.12111395. No abstract available. PMID 23820835
- [Derived] Mason AE, Chowdhary A, Hartogensis W, Siwik CJ, Lupesko-Persky O, Pandya LS, Roberts S, Anglo C, Moran PJ, Nelson JC, Lowry CA, Patrick RP, Raison CL, Hecht FM. Feasibility and acceptability of an integrated mind-body intervention for depression: whole-body hyperthermia (WBH) and cognitive behavioral therapy (CBT). Int J Hyperthermia. 2024;41(1):2351459. doi: 10.1080/02656736.2024.2351459. Epub 2024 May 14. PMID 38743265
- See also: Access to initial online screening for interested prospective participants — https://www.sealab.ucsf.edu/heatbedstudy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.47 (13.89) | 35.87 (13.06) | 38.17 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Latino/Hispanic | 5 | 4 | 9
  White/Caucasian | 7 | 4 | 11
  More than one race | 1 | 2 | 3
  Unreported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Education (highest level completed) [Count of Participants; unit: Participants]
  High School diploma or GED | 0 | 0 | 0
  Some college | 1 | 1 | 2
  Associate's Degree | 1 | 3 | 4
  Bachelor's Degree | 8 | 5 | 13
  Master's Degree | 5 | 3 | 8
  Professional Degree (e.g., MD, DDS, JD) | 0 | 1 | 1
  Doctoral Degree (e.g., PhD, EdD) | 0 | 2 | 2
Body Mass Index (BMI), Kg/m^2 [Mean (Standard Deviation); unit: kg/m^2 (kilograms per meter-squared)] | 27.12 (6.45) | 25.93 (5.54) | 26.53 (5.94)
Blood Pressure (SBP/DBP), mm Hg [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure | 114.2 (14.2) | 113.0 (17.2) | 113.6 (15.5)
  Diastolic Blood Pressure | 76.3 (8.6) | 78.7 (8.6) | 77.5 (8.5)
Beck Depression Inventory II (BDI-II) [Mean (Standard Deviation); unit: Score on a scale] — Scores range from 0 to 63 and items are summed to create a total score; higher scores indicate greater depression symptoms.
  Score on a scale | 32.73 (9.07) | 32.27 (7.76) | 32.50 (8.30)

OUTCOME MEASURES:

1. Primary Outcome: Net Promoter Score, and Enrollment Likelihood
Description: Study acceptability was indexed by participant-reported net-promoter scores. This is a response to a single question: "How likely would you be to recommend [participation in a study or treatment like this] to a friend or family member with depression?" Net promoter scores range from 0 (would not recommend) to 10 (would definitely recommend). Study acceptability was also indexed by an additional patient-reported metric, Enrollment Likelihood. Enrollment likelihood was a response to the question: "How likely would you be to enroll in this study given your experience in this study?" and response options range from 1 (extremely unlikely) to 5 (extremely likely).
Time Frame: 12 weeks
Population: Study participants who completed the final study survey, Net Promoter Score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
Number analyzed (Participants) | 15 | 14
score on a scale
  Net Promoter Score (0-10) | 7.73 (2.15) | 8.00 (2.08)
  Enrollment Likelihood (1-5) | 4.13 (1.06) | 4.29 (0.83)

2. Secondary Outcome: Change in Beck Depression Inventory-II (BDI-II)
Description: Change in BDI-II from baseline assessment to final assessment. Scores range from 0 to 63 and items are summed to create a total score; higher scores indicate greater depression symptoms.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
Number analyzed (Participants) | 15 | 14
score on a scale | -19.07 (2.69) | -21.10 (2.41)

3. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS) 8a Depression
Description: Change in PROMIS8a Depression from baseline to final assessment. T scores are computed; higher scores indicate greater depression symptoms. A T-score of 60 indicates sub-clinical or elevated levels of depression. A T score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: T-score units
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
Number analyzed (Participants) | 15 | 14
T-score units | -10.79 (2.66) | -11.54 (2.84)

4. Secondary Outcome: Change in Hamilton Depression Rating Scale 6-item (HAMD-6) Self-Report
Description: Change in HAMD-6 from baseline to final assessment. Scores range from 0 to 22, and items are summed to create a total score; higher scores indicate greater depression symptoms.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
Number analyzed (Participants) | 15 | 14
score on a scale | -6.42 (1.30) | -7.16 (1.12)

5. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information Systems (PROMIS) 4a Anxiety
Description: Change in PROMIS4a Anxiety from baseline to final assessment. T scores are computed; higher scores indicate greater depression symptoms. A T-score of 60 indicates sub-clinical or elevated levels of anxiety. A T score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: T-score units
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
Number analyzed (Participants) | 15 | 14
T-score units | -7.24 (1.63) | -7.51 (2.06)

6. Other Pre Specified Outcome: Sudden Gains in Antidepressant Responses
Description: Sudden gain in BDI-II scores, defined as >25% reduction in depression symptoms in between between two adjacent sauna sessions, account for more than 50% of total depression symptom improvement
Time Frame: 2-3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active Whole-body Hyperthermia (Active Treatment) | Sham Whole-body Hyperthermia (Sham Treatment)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 14/15 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Whole-body Hyperthermia (Active Treatment) (N=15) | Sham Whole-body Hyperthermia (Sham Treatment) (N=15)
Headache (Nervous system disorders) | 13 (28) | 3 (6) — Headache
Lightheadedness (General disorders) | 7 (15) | 2 (3) — Lightheadedness
Migraine (Nervous system disorders) | 1 (2) | 0 (0) — Migraine
Nausea (Gastrointestinal disorders) | 5 (8) | 2 (2) — Nausea
Fatigue (General disorders) | 1 (2) | 0 (0) — Fatigue
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Emesis
Bruising (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Bruising
Sleep Disturbance (General disorders) | 1 (1) | 0 (0) — Sleep Disturbance
Head Pressure (General disorders) | 1 (1) | 0 (0) — Head Pressure
Chills (General disorders) | 1 (1) | 0 (0) — Chills
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Stomach pain
Dry mouth (General disorders) | 1 (1) | 0 (0) — Dry mouth
Flu (Infections and infestations) | 0 (0) | 1 (1) — Flu
Knee surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Knee surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT05708976/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT05708976/ICF_001.pdf